CLINICAL TRIAL: NCT06667700
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Clinical Study to Evaluate the Efficacy and Safety of Molnupiravir (MK-4482) in Non-Hospitalized Adults With COVID-19 at High Risk for Disease Progression
Brief Title: A Clinical Study of Molnupiravir to Prevent Severe Illness From Coronavirus Disease 2019 (COVID-19) in People Who Are High Risk (MK-4482-023)
Acronym: MOVe-NOW
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4482-023; 2023-507227-36-00 (Registry Identifier: EU CT); U1111-1295-4678 (Registry Identifier: UTN); MK-4482-023 (Other: MSD); jRCT2031250022 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Molnupiravir (Experimental): Participants will receive 800 mg molnupiravir orally every 12 hours for 5 days (a total of 10 consecutive doses)
  Interventions: Drug: Molnupiravir
- Placebo (Placebo Comparator): Participants will receive molnupiravir-matching placebo orally every 12 hours for 5 days (a total of 10 consecutive doses)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Molnupiravir — Molnupiravir administered orally as two 400 mg film-coated tablets every 12 hours for 5 days (a total of 10 consecutive doses)
  Other Names: MK-4482; LAGEVRIO®
  Arms: Molnupiravir
Drug: Placebo — Molnupiravir-matching placebo administered orally as two film-coated tablets every 12 hours for 5 days (a total of 10 consecutive doses)
  Arms: Placebo

SUMMARY:
Researchers are looking for other ways to prevent severe illness from COVID-19. COVID-19 is a virus that most often causes mild flu or cold-like symptoms. However, people with certain health conditions or other factors have a high risk (chance) of getting severely ill from COVID-19, which can require a hospital stay or lead to death. Some people who are high risk for severe illness may be unable to take certain treatments for COVID-19 because they are not available to them, or they take other medicines that may react with a treatment and cause an unwanted effect.

Molnupiravir (MK-4482) is a study medicine designed to stop the COVID-19 virus from copying itself in the body (multiplying). The goal of this study is to learn if molnupiravir prevents severe illness from COVID-19 more than placebo in people who are high risk.

ELIGIBILITY:
Inclusion Criteria

The main inclusion criteria include but are not limited to the following:

* Is an individual of any sex/gender, ≥18 years of age
* Has documentation of SARS-CoV-2 infection with sample collection ≤4 days prior to randomization
* Has initial onset of signs/symptoms attributable to COVID-19 for ≤4 days prior to the day of randomization and ≥2 of the following signs/symptoms attributable to COVID-19 on the day of randomization: cough, sore throat, nasal congestion, shortness of breath or difficulty breathing with exertion, muscle or body aches, fatigue, fever >38.0°C or chills, nausea or vomiting or diarrhea, change in sense of smell or change in sense of taste, or headache
* Has ≥1 of the following characteristics or medical conditions associated with the highest risk of severe illness from COVID-19:

  * Advanced age of ≥75 years of age
  * Immunocompromised
  * Neurocognitive or physical disability
  * Has ≥3 characteristics or medical conditions which increase the risk of severe illness due to COVID-19 (e.g., chronic lung disease, obesity with body mass index (BMI) ≥35, diabetes)
* Is unable or unwilling to receive treatment with nirmatrelvir/ritonavir (NMV/r) due to 1 or more of the following:

  * Is receiving drug(s) highly dependent on cytochrome P450 3A (CYP3A) for clearance and for which elevated concentrations are associated with serious and/or life-threatening consequences or drug(s) with a clinically significant drug-drug interaction for which co-administration is not possible
  * Is receiving potent CYP3A inducers where significantly reduced nirmatrelvir or ritonavir plasma concentrations may be associated with the potential for loss of virologic response and possible resistance
  * Has severe hepatic impairment
  * Has experienced prior adverse reactions or hepatotoxicity to NMV/r that would preclude future use
  * Has known or suspected NMV/r resistance
  * Has uncontrolled HIV infection
  * NMV/r is not approved/authorized in the participant's country or it is not accessible to participant (e.g., drug shortage)
  * Is unwilling to receive treatment with NMV/r

Inclusion note: Participants may receive remdesivir as standard of care in addition to molnupiravir or placebo. If remdesivir is available and clinically appropriate per local clinical practice, investigators will aim to ensure that those who are most vulnerable to severe COVID-19 receive timely access to remdesivir as standard of care on this study.

Exclusion Criteria

The main exclusion criteria include but are not limited to the following:

* Is currently hospitalized or is expected to need hospitalization for COVID-19 imminently
* Has received or plans to receive SARS-CoV-2 directed oral antivirals or monoclonal antibodies for current episode of COVID-19 (other than study intervention and, if applicable, remdesivir as standard of care)
* Has ≥1 of the following signs/symptoms that are attributable to severe or critical COVID-19:

  * Shortness of breath at rest
  * Respiratory rate ≥30 breaths per minute
  * Heart rate ≥125 beats per minute
  * Peripheral oxygen saturation (SpO2) ≤93% on room air or on supplemental oxygen for a reason other than COVID-19 which has not increased since onset of COVID-19 signs/symptoms
  * New or increasing need for supplemental oxygen: receiving >4 liters/minute supplemental oxygen due to COVID-19 OR on supplemental oxygen for a reason other than COVID-19 which has increased due to COVID-19
* Has received a COVID-19 vaccine within 30 days prior to randomization
* Has a history of confirmed influenza, respiratory syncytial virus (RSV), or SARS-CoV-2 infection (with or without symptoms; excluding current infection) within 30 days prior to randomization
* Has known or suspected hypersensitivity to active or inactive ingredients of molnupiravir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3082 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2031-01-26 (Estimated); Study Completion 2031-01-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced One or More of Following Through Day 29: All-cause Hospitalization, All-cause Mortality, or Covid-19-related Medically-attended Visit (MAV) | Up to 29 days
  Hospitalization is defined as ≥24 hours of acute care in a hospital or similar acute care facility, including emergency rooms or facilities created to address hospitalization needs specifically for COVID-19. Hospitalization and death may be due to any cause. An MAV is defined as any unscheduled, nonroutine healthcare visit where the participant is evaluated by a licensed (according to local/national guidelines) healthcare provider. As prespecified by the protocol, the percentage of participants who experience ONE OR MORE of these 3 events (hospitalization, death, or COVID-19-related MAV) occurring from randomization through Day 29 will be presented.
Percentage of Participants Who Experienced an Adverse Event (AE) | Up to approximately 5 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with at least 1 AE will be presented.
Percentage of Participants Who Discontinued Study Intervention Due to AE | Up to approximately 5 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study intervention due to an AE will be presented.

SECONDARY OUTCOMES:
Time to Sustained Alleviation (without relapse) of all selected 8 (5 prespecified and 3 determined by baseline prevalence), self-reported COVID-19 signs/symptoms | Up to 29 days
  Time to sustained alleviation without relapse is defined as the number of days from randomization to the first of 2 consecutive days when alleviation (lessening of symptoms) is demonstrated, collectively, for all 8 selected COVID-19-related sign/symptoms. Participants who experience sustained alleviation for 2 consecutive days must not relapse in any of the 8 signs/symptoms before Day 29. The time to sustained alleviation without relapse of all 8 selected COVID-19-related signs/symptoms from randomization through Day 29 will be presented.
Change from Baseline in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) RNA Titer | Day 1 (baseline) and up to Day 29
  SARS-CoV-2 RNA titer (viral load) will be measured by quantitative reverse transcriptase polymerase chain reaction (RT-PCR) of samples from nasopharyngeal (NP) swabs, and the mean change from baseline will be presented.
Percentage of Participants with Undetectable SARS-CoV-2 RNA | Up to 29 days
  SARS-CoV-2 RNA (viral load) will be measured by quantitative RT-PCR of samples from NP swabs, and the percentage of participants with undetectable (i.e., below the lower limit of quantification) SARS-CoV-2 RNA (viral load) will be presented.
Percentage of Participants Who Experienced One or More of Following Through Day 29: All-cause Hospitalization or All-cause Mortality | Up to 29 days
  Hospitalization is defined as ≥24 hours of acute care in a hospital or similar acute care facility, including emergency rooms or facilities created to address hospitalization needs specifically for COVID-19. Hospitalization and death may be due to any cause. As prespecified by the protocol, the percentage of participants who experience hospitalization AND/OR death occurring from randomization through Day 29 will be presented.
Percentage of Participants With Clinically Important Medical Interventions (CIMI) Associated with COVID-19-related MAV or COVID-19-related Hospitalization Through Day 29 | Up to 29 days
  CIMIs were prespecified by the protocol and include, but are not limited to, supplemental oxygen therapy, IV fluid administration, and nebulizer treatment. An MAV is defined as any unscheduled, nonroutine healthcare visit where the participant is evaluated by a licensed (according to local/national guidelines) healthcare provider. Hospitalization is defined as ≥24 hours of acute care in a hospital or similar acute care facility, including emergency rooms or facilities created to address hospitalization needs specifically for COVID-19. The percentage of participants with CIMIs associated with a COVID-19-related MAV AND/OR a COVID-19-related hospitalization through Day 29 will be reported.
Time to Sustained Alleviation (without relapse) of all 15 self-reported COVID-19 signs/symptoms through Day 29 | Up to 29 days
  Time to sustained alleviation without relapse is defined as the number of days from randomization to the first of 2 consecutive days when alleviation (lessening of symptoms) is demonstrated, collectively, for all 15 COVID-19-related sign/symptoms. Participants who experience sustained alleviation after 2 consecutive days must not relapse in any of the 15 signs/symptoms before Day 29. The time to sustained alleviation without relapse of all 15 COVID-19-related signs/symptoms from randomization through Day 29 will be presented.
Time to Sustained Resolution Without Relapse of all 8 (5 prespecified and 3 determined by baseline prevalence) self-reported COVID-19 signs/symptoms through Day 29 | Up to 29 days
  Time to sustained resolution without relapse is defined as the number of days from randomization to the first of 2 consecutive days when resolution (having no symptoms or only mild symptoms) is demonstrated, collectively, for all 8 selected COVID-19-related sign/symptoms. Participants who experience sustained resolution after 2 consecutive days must not relapse in any of the 8 signs/symptoms before Day 29. The time to sustained resolution without relapse of all 8 selected COVID-19-related signs/symptoms from randomization through Day 29 will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (215):
- United States (71):
  - Cullman Clinical Trials ( Site 3813), Cullman, Alabama
  - Helios Clinical Research ( Site 3826), Paradise Valley, Arizona
  - Absolute Clinical Research ( Site 3709), Phoenix, Arizona
  - Clinica de Salud del Valle de Salinas ( Site 3825), Castroville, California
  - Ascada Health PC dba Ascada Research ( Site 3750), Fullerton, California
  - Pacific Clinical Studies ( Site 3827), Los Alamitos, California
  - Valley Clinical Trials, Inc. ( Site 3707), Northridge, California
  - FOMAT Medical Research ( Site 3720), Oxnard, California
  - Paradigm Clinical Research, LLC ( Site 3785), San Diego, California
  - Optimus Medical ( Site 3817), San Francisco, California
  - Millennium Clinical Trials ( Site 3758), Westlake Village, California
  - Paradigm Clinical Research Centers, Inc ( Site 3718), Wheat Ridge, Colorado
  - Encore Medical Research of Boynton Beach ( Site 3701), Boynton Beach, Florida
  - Prestige Clinical Research Center ( Site 3722), Coral Gables, Florida
  - Indago Research & Health Center, Inc ( Site 3714), Hialeah, Florida
  - Prestige Clinical Research ( Site 3830), Homestead, Florida
  - Accel Research Sites Network - St. Pete-Largo Clinical Research Unit ( Site 3779), Largo, Florida
  - Clinical Site Partners, LLC dba Flourish Research ( Site 3717), Leesburg, Florida
  - Advanced Pulmonary Research Institute ( Site 3781), Loxahatchee Groves, Florida
  - Southern Clinical Research ( Site 3773), Miami, Florida
  - Florida Pharmaceutical Research and Associates ( Site 3763), Miami, Florida
  - Bio-Medical Research LLC ( Site 3804), Miami, Florida
  - Bright Research Center ( Site 3746), Miami, Florida
  - Miami Clinical Research ( Site 3729), Miami, Florida
  - Reed Medical Research ( Site 3761), Miami, Florida
  - Palm Springs Community Health Center ( Site 3757), Miami Lakes, Florida
  - Panax Clinical Research ( Site 3803), Miami Lakes, Florida
  - Combined Research Orlando Phase I-IV ( Site 3797), Orlando, Florida
  - CDC Research Institute ( Site 3716), Port Saint Lucie, Florida
  - New Tampa Health ( Site 3764), Tampa, Florida
  - Clinical Research Trials of Florida ( Site 3703), Tampa, Florida
  - Precision Research Center ( Site 3704), Tampa, Florida
  - Encore Medical Research - Weston ( Site 3708), Weston, Florida
  - Balanced Life Health Care Solutions/SKYCRNG ( Site 3713), Lawrenceville, Georgia
  - Renew Health Clinical Research ( Site 3760), Snellville, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG ( Site 3816), Union City, Georgia
  - Paradigm Clinical Research - Boise ( Site 3841), Boise, Idaho
  - Rush University Medical Center ( Site 3748), Chicago, Illinois
  - Duly Health and Care ( Site 3799), Lombard, Illinois
  - University of Louisville School of Medicine ( Site 3706), Louisville, Kentucky
  - Barnum Medical Research ( Site 3828), Natchitoches, Louisiana
  - Annapolis Internal Medicine - CCT Research ( Site 3700), Annapolis, Maryland
  - Kur Research - Columbia Medical ( Site 3767), Columbia, Maryland
  - Revival Research Institute, LLC ( Site 3835), Dearborn, Michigan
  - Michigan Center of Medical Research (MICHMER) ( Site 3734), Farmington Hills, Michigan
  - Henry Ford St John TM Center for Infectious Disease Research ( Site 3766), Grosse Pointe Woods, Michigan
  - Mankato Clinic ( Site 3842), Mankato, Minnesota
  - Prime Health and Wellness/SKYCRNG ( Site 3726), Fayette, Mississippi
  - SKY Integrative Medical Center/SKYCRNG ( Site 3740), Ridgeland, Mississippi
  - Nevada Health Centers ( Site 3840), Carson City, Nevada
  - WR-CRCN, LLC ( Site 3818), Las Vegas, Nevada
  - Saint Michael's Medical Center ( Site 3808), Newark, New Jersey
  - Holy Name Medical Center ( Site 3807), Teaneck, New Jersey
  - Weill Cornell Medical College ( Site 3814), New York, New York
  - Prime Global Research ( Site 3731), The Bronx, New York
  - OnSite Clinical Solutions ( Site 3784), Charlotte, North Carolina
  - Monroe Biomedical Research ( Site 3732), Monroe, North Carolina
  - IMA Clinical Research Mount Airy ( Site 3745), Mount Airy, North Carolina
  - Research Innovations, LLC ( Site 3712), Beavercreek, Ohio
  - Midlands Neurology & Pain Associates ( Site 3751), Columbia, South Carolina
  - Helios Clinical Research - JAC ( Site 3833), Jackson, Tennessee
  - Javara - Privia Medical Group Gulf Coast - The Woodlands HWH ( Site 3837), Conroe, Texas
  - South Texas Clinical Research ( Site 3815), Corpus Christi, Texas
  - Care United Research, LLC ( Site 3747), Forney, Texas
  - Houston Methodist Hospital ( Site 3800), Houston, Texas
  - MD Anderson ( Site 3843), Houston, Texas
  - Andres Garcia Zuniga, M.D., P.A. ( Site 3782), Laredo, Texas
  - LinQ Research ( Site 3824), Pearland, Texas
  - Crossroads Clinical Research-Family Practice ( Site 3739), Victoria, Texas
  - Velocity Clinical Research - Hampton ( Site 3744), Hampton, Virginia
  - Eastside Research Associates ( Site 3727), Redmond, Washington
- Argentina (4):
  - CEMIC ( Site 0101), Buenos Aires., Buenos Aires
  - Hospital Italiano de Buenos Aires ( Site 0107), Ciudad Autonoma de Buenos Aires., Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0111), Mar del Plata, Buenos Aires
  - Nefra Medical Care - Moron ( Site 0109), Morón, Buenos Aires
- Brazil (3):
  - Hospital Felicio Rocho (HFR) - Nucleo de Ciencias da Saude ( Site 0402), Belo Horizonte, Minas Gerais
  - Centro de Pesquisa Sao Lucas ( Site 0401), Campinas, São Paulo
  - Centro de Pesquisa Clinica Institucional do HCFMUSP - CPCi ( Site 0403), São Paulo
- Bulgaria (10):
  - Medical Center Asclepius ( Site 0506), Velingrad, Pazardzhik
  - Medical Center Zdrave 1 ( Site 0509), Kozloduy, Vratsa
  - Medconsult Pleven - Lovech ( Site 0501), Lovech
  - Medical Center Hera ( Site 0507), Montana
  - MHAT "Dr. Stamen Iliev" Montana-Department of Pulmonology ( Site 0504), Montana
  - Medconsult Pleven ( Site 0503), Pleven
  - DKC V - Plovdiv ( Site 0508), Plovdiv
  - SHATPPD Dr. Dimitar Gramatikov - Ruse EOOD ( Site 0502), Rousse
  - Diagnostic Consultative Center 22 - Sofia ( Site 0500), Sofia
  - Medical Center Hera EOOD ( Site 0505), Sofia
- Colombia (7):
  - IPS SURA San Diego ( Site 0806), Medellín, Antioquia
  - IPS Centro Científico Asistencial S.A.S ( Site 0800), Barranquilla, Atlántico
  - Clinica Colsanitas - Sede Reina Sofia ( Site 0807), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 0804), Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS-Oncology ( Site 0801), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 0805), Montería, Departamento de Córdoba
  - Fundación Valle del Lili ( Site 0803), Cali, Valle del Cauca Department
- MeVac - Meilahti Vaccine Research Center ( Site 1200), Helsinki, Uusimaa, Finland
- France (4):
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital F-Centre d'Investigation Clinique - Plur ( Site 1301), Dijon, Bourgogne-Franche-Comté
  - CHU de Saint-Etienne ( Site 1302), Saint Priest En Jarez, Pays de la Loire Region
  - centre hospitalier lyon sud ( Site 1303), Pierre-Bénite, Rhone
  - Pitie Salpetriere University Hospital-Infectious Disease - Tropical Diseases ( Site 1300), Paris, Île-de-France Region
- Georgia (8):
  - Clinic Health - Batumi ( Site 1405), Batumi, Adjara
  - Family Medical Regional Center ( Site 1404), Batumi, Adjara
  - LTD High Technology Hospital Medcenter ( Site 1408), Batumi, Adjara
  - University Clinic of Innovative Medicine ( Site 1400), Batumi, Adjara
  - Caucasus Medical Centre ( Site 1406), Tbilisi, Adjara
  - "Georgian Clinics" JSC ( Site 1410), Zugdidi, Samegrelo and Zemo Svaneti
  - New Hospitals ( Site 1409), Tbilisi
  - Curatio Clinic - Main Location ( Site 1401), Tbilisi
- Germany (4):
  - TUM Klinikum ( Site 1502), Munich, Bavaria
  - Universitätsklinikum Frankfurt Goethe-Universität ( Site 1503), Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln ( Site 1505), Cologne, North Rhine-Westphalia
  - Campus Charite Mitte Nephrologie und Internistische Intensivmedizin ( Site 1501), Berlin, State of Berlin
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 1904), Bologna
  - Ospedale San Martino ( Site 1900), Genova
  - ASST Fatebenefratelli Sacco ( Site 1901), Milan
  - AOU Pisana- Ospedale Cisanello ( Site 1905), Pisa
- Japan (6):
  - National Hospital Organization Shimoshizu National Hospital ( Site 2007), Yotsukaidō, Chiba
  - Tsuchiura Beryl Clinic ( Site 2009), Tsuchiura, Ibaraki
  - National Hospital Organization Tokyo National Hospital ( Site 2003), Kiyose, Tokyo
  - Sekino Hospital ( Site 2016), Toshimaku, Tokyo
  - National Hospital Organization Kyushu Medical Center ( Site 2006), Fukuoka
  - Kumamoto Chuo Hospital ( Site 2002), Kumamoto
- Mexico (8):
  - Morales Vargas Centro de Investigacion ( Site 2206), León, Guanajuato
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 2207), Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran-Departamento de Infectología ( Site 2203), Mexico City, Mexico City
  - Instituto Nacional de Salud Publica ( Site 2205), Cuernavaca, Morelos
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Infectologia ( Site 2204), Monterrey, Nuevo León
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan ( Site 2202), Mérida, Yucatán
  - ICARO Investigaciones en Medicina ( Site 2200), Chihuahua City
  - Arké SMO S.A de C.V-ARKE SMO S.A. de C.V. ( Site 2210), Veracruz
- New Zealand (8):
  - CGM Research Trust ( Site 2307), Christchurch, Canterbury
  - Pacific Clinical Research Network - Tasman ( Site 2304), Nelson, Tasman District
  - Lakeland Clinical Trials Waikato ( Site 2302), Nawton, Waikato Region
  - Lakeland Clinical Trials Wellington ( Site 2303), Upper Hutt, Wellington Region
  - Pacific Clinical Research Network West Auckland ( Site 2301), Auckland
  - Optimal Clinical Trials North ( Site 2308), Auckland
  - Silverdale Medical Limited ( Site 2305), Auckland
  - Optimal Clinical Trials ( Site 2306), Auckland
- Peru (2):
  - Asociación Civil Selva Amazónica ( Site 2405), Iquitos, Loreto
  - Clinica Ricardo Palma-Centro de Investigacion de Enfermedades Respiratorias Thorax ( Site 2404), Lima
- Philippines (2):
  - Health Index Multispeciality Clinic ( Site 2501), Bacoor, Cavite
  - GreenCity Medical Center ( Site 2503), San Fernando City, Pampanga
- Poland (7):
  - PL Certus ( Site 2613), Poznan, Greater Poland Voivodeship
  - In-Vivo Bydgoszcz ( Site 2601), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - NZOZ GynCentrum - Oddział Kraków ( Site 2609), Krakow, Lesser Poland Voivodeship
  - Penta Hospitals Przychodnie Wrocław Wejherowska ( Site 2611), Wroclaw, Lower Silesian Voivodeship
  - NZOZ GynCentrum - Oddział Bielsko-Biała ( Site 2602), Bielsko-Biala, Silesian Voivodeship
  - Clinical Medical Research ( Site 2604), Katowice, Silesian Voivodeship
  - Holsamed ( Site 2603), Katowice, Silesian Voivodeship
- Puerto Rico (3):
  - Investigadores del Este LLC ( Site 4001), Humacao
  - Miralles Clinical Research LLC ( Site 4004), San Juan
  - MV HEALTH SERVICES LLC ( Site 4003), San Juan
- Romania (6):
  - Spitalul Clinic de Boli Infecțioase și Tropicale Victor Babeș ( Site 2701), Bucharest, București
  - Spitalul Clinic De Urgenta Prof Dr Agrippa Ionescu ( Site 2705), Baloteşti, Ilfov
  - Centrul Medical SANA ( Site 2704), Bucharest
  - National Institute for Infectious Diseases Prof. Dr. Matei Bals ( Site 2706), Bucharest
  - Spitalul Clinic de Boli Infecțioase ( Site 2703), Cluj-Napoca
  - Spitalul Clinic de Boli Infecțioase ( Site 2702), Constanța
- South Korea (9):
  - Wonju Severance Christian Hospital-Internal Medicine ( Site 3009), Wŏnju, Kang-won-do
  - Chonnam National University Hospital-Infectious Diseases ( Site 3008), Gwangju, Kwangju-Kwangyokshi
  - Korea University Ansan Hospital ( Site 3007), Ansan-si, Kyonggi-do
  - Gyeongsang National University Hospital ( Site 3005), Jinju, Kyongsangnam-do
  - Pusan National University Hospital-Internal Medicine ( Site 3010), Pusan, Pusan-Kwangyokshi
  - Kyungpook National University Chilgok Hospital-Division of Infectious Diseases ( Site 3002), Deagu, Taegu-Kwangyokshi
  - Korea University Anam Hospital ( Site 3001), Seoul
  - Hallym University Kangnam Sacred Heart Hospital-Internal Medicine ( Site 3003), Seoul
  - Korea University Guro Hospital ( Site 3006), Seoul
- Spain (9):
  - Hospital General Universitario de Elche-Infectius Disease ( Site 3105), Elche, Alicante
  - Hospital Germans Trias i Pujol ( Site 3101), Badalona, Barcelona
  - EAP Osona Sud - Alt Congost S.L.P ( Site 3107), Centelles, Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 3102), Barcelona, Catalonia
  - Hospital Universitario de A Coruña ( Site 3112), A Coruña, Galicia
  - Hospital Santa Lucia-Medicina Infecciosas ( Site 3106), Cartagena, Murcia
  - EAP Sardenya ( Site 3109), Barcelona
  - Hospital Universitario Infanta Leonor ( Site 3110), Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO ( Site 3100), Seville
- Taiwan (9):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 3306), Kaoshiung, Kaohsiung
  - Taoyuan General Hospital ( Site 3300), Taoyuan, Taoyuan
  - Kaohsiung Veterans General Hospital ( Site 3307), Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital ( Site 3308), New Taipei City
  - Taichung Veterans General Hospital ( Site 3305), Taichung
  - National Taiwan University Hospital ( Site 3301), Taipei
  - Tri-Service General Hospital ( Site 3304), Taipei
  - Taipei Municipal Wangfang Hospital ( Site 3309), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 3303), Taoyuan District
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital-Department of Medicine ( Site 3401), Bangkok, Bangkok
  - HIV Netherlands Australia Thailand Research Collaboration ( Site 3402), Pathumwan, Bangkok
- Ukraine (19):
  - EUROMEDCLINIC ( Site 3517), Cherkasy, Cherkasy Oblast
  - MUNICIPAL NON-PROFIT ENTERPRISE CENTRAL CITY CLINICAL HOSPITAL OF CHERNIVTSI CITY COUNCIL ( Site 3513), Chernivtsi, Chernihiv Oblast
  - Clinical medical and diagnostic center Limited Liability Company "Simedgroup" ( Site 3524), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Regional Phthisiology and Pulmonology Center ( Site 3523), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Private Enterprise Private Manufacturing Company Acinus-Medical and Diagnostic Centre ( Site 3537), Kropyvnytskyi, Kirovohrad Oblast
  - Limited Liability Company Ukrainian Center of Tomotherapy-Clinical Trials Department ( Site 3512), Kropyvnytskyi, Kirovohrad Oblast
  - Medical Center "Harmoniya Krasy" ( Site 3545), Kyiv, Kyivska Oblast
  - Edelweiss Medics ( Site 3503), Kyiv, Kyivska Oblast
  - Communal Non-Profit Enterprise "Kyiv City Clinical Hospital #1"-Department of Clinical Research ( Site 3514), Kyiv, Kyivska Oblast
  - Medbud Clinic-Treatment prevention unit ( Site 3506), Kyiv, Kyivska Oblast
  - Medical Center of Limited ( Site 3546), Kyiv, Kyivska Oblast
  - Center of Family Medicine Plus ( Site 3502), Kyiv, Kyivska Oblast
  - Polyclinic of Communal 4th city clinical hospital ( Site 3501), Lviv, Lviv Oblast
  - University clinic of the National Pirogov Memorial Medical University ( Site 3547), Vinnytsia, Vinnytsia Oblast
  - Clinic of Pyrohov National Medical University of Vinnytsia ( Site 3528), Vinnytsia, Vinnytsia Oblast
  - Municipal Enterprise "Volyn Regional Clinical Hospital" of Volyn Regional Council ( Site 3530), Lutsk, Volyn Oblast
  - Uzhhorod Municipal Multidisciplinary Clinical Hospital of Uzhhorod City Council ( Site 3538), Uzhhorod, Zakarpattia Oblast
  - Medlight Clinic ( Site 3548), Kyiv
  - Kyiv Railway Clinical Hospital No.2 of Branch Health Center -Center of Clinical Trials ( Site 3549), Kyiv
- United Kingdom (9):
  - Whiteladies Medical Group ( Site 3611), Bristol, Bristol, City of
  - Royal Devon & Exeter Hospital ( Site 3604), Exeter, England
  - Royal Victoria Infirmary ( Site 3608), Newcastle, Newcastle Upon Tyne
  - Norwich Practices Health Centre ( Site 3605), Norwich, Norfolk
  - Oak Street Medical Practice ( Site 3612), Norwich, Norfolk
  - Lakeside Surgery ( Site 3600), Northamptonshire, Northamptonshire
  - Bicester Health Centre ( Site 3609), Bicester, Oxfordshire
  - Banbury Cross Health Centre ( Site 3610), Oxford, Oxfordshire
  - Buttercross Health Centre ( Site 3606), Somerset, Somerset

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Protocol Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26184&tenant=MT_MSD_9011